CLINICAL TRIAL: NCT00027391
Title: Clinical Trials of Albuterol and Oxandrolone in FSH Dystrophy
Brief Title: Study of Albuterol and Oxandrolone in Patients With Facioscapulohumeral Dystrophy (FSHD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FDA Office of Orphan Products Development (U.S. Federal Agency)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: FD-R-2029-01; FD-R-002029-01
Record Dates: First submitted 2001-12-05; First posted 2001-12-07 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2001-11

CONDITIONS: Muscular Dystrophies
Keywords: Muscle Weakness, Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophies; Muscle Weakness | interventions — Albuterol; Oxandrolone

INTERVENTIONS:
Drug: Albuterol
Drug: Oxandrolone

SUMMARY:
This is a study to determine whether albuterol or oxandrolone, alone or in combination, are able to increase strength and muscle mass in patients with FSHD. It also will determine if albuterol given in "pulsed" fashion will have more effect than when given continuously.

DETAILED DESCRIPTION:
Patients will be randomized to 1 of 4 groups: placebo, pulsed albuterol, oxandrolone, or both pulsed albuterol and oxandrolone. Treatment will continue for 52 weeks unless unacceptable side effects occur. Patients will undergo testing of muscle function. All patients will return for follow-up assessments at Weeks 4, 12, 26, and 52.

ELIGIBILITY:
Inclusion criteria:

* Presence of 4q35 "small fragment" of less than 40 kb by standard DNA testing
* Weakness of the facial muscles, including frontalis, orbicularis oculi, or orbicularis oris
* Weakness of scapular stabilizers or foot dorsiflexors
* Ambulatory
* Weakness grade 2 or worse in the arm using upper extremity grading scale

Exclusion criteria:

* Prior use of oral beta-2 agonists for a period of at least 1 year or within the past 3 months
* Concurrent use of other sympathomimetic agents, antidepressants, or beta-2 receptor blockers
* Pregnancy
* Known hypersensitivity to anabolic steroids
* Any medical or psychological condition that would interfere with the study
* Requirement for a wheelchair

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160
Dates: Start 2001-09; Study Completion 2004-08

CONTACTS AND LOCATIONS:
Overall Officials: John T. Kissel, M.D., Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States